CLINICAL TRIAL: NCT04615104
Title: Functional, Clinical, and Performance Outcomes Following Pelvic and Acetabular Fracture: A Prospective Observational Study
Brief Title: Pelvic and Acetabular Fracture: A Prospective Observational Study
Acronym: PACE
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00082574; 10-19-18E (Other: Atrium)
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Fracture; Acetabular Fracture; Pubic Rami Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pelvic Ring Fracture: Patients with pelvic ring fractures.
  Interventions: Procedure: Operative; Procedure: Nonoperative
- Acetabular Fracture: Patients with acetabular fractures.
  Interventions: Procedure: Operative; Procedure: Nonoperative

INTERVENTIONS:
Procedure: Operative — surgical treatment
Procedure: Nonoperative — nonsurgical treatment

SUMMARY:
The purpose of this study is to understand the trajectory of function and self-reported outcomes of patients following pelvic and acetabular, treated both operatively and nonoperatively.

DETAILED DESCRIPTION:
The goal of the study study is to prospectively capture data from patients following pelvic and acetabular fractures, treated both operatively and nonoperatively, in order to understand the trajectory of functional and self-reported outcomes as well as to answer critical questions about treatment. Performance assessment data and patient-reported outcome measures utilizing the NIH PROMIS tool will be collected and analyzed for patients following pelvic or acetabular fracture, regardless of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the pelvic ring
* Fracture of the acetabulum

Exclusion Criteria:

* Patients unwilling to provide consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for pelvic or acetabular fracture at an orthopaedic trauma practices.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Return to work/activities | 0-24 months following injury
  Average time to return to work and activities

SECONDARY OUTCOMES:
Change in patient-reported outcomes measurement information system (PROMIS 29) scores | baseline, 3, 6, 12 and 24 months
  The PROMIS-29 assesses seven health domains: physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and ability to participate in social roles and activities. Each of the seven domains has four questions which are scored on a five-point Likert scale. The PROMIS-29 scales will be scored using a T-score metric method available at the Assessment Center website (http://assessmentcenter.net). A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores mean more of the specific scale's construct, which may indicate a desirable or an undesirable outcome.
Fracture Healing | 0-24 months following injury
  Union rates as measured clinically and radiographically. Xrays will be collected from the electronic medical record.
Complications | 0-24 months following injury
  Rates of readmission, reoperations and complications
Performance Measure- 10 meter walk test | 3, 6, 12 and 24 months
  Participants complete a modified 10 meter walk test which involves the subject starting from a standing position, walking 5 meters at a comfortable pace, turning around, and then walking back 5 meters to the original starting point. The test is repeated twice for each subject.
Performance Measure- Five Time Sit to Stand Test | 3, 6, 12 and 24 months
  Participants begin from a seated position and are directed to come to a full standing position without push off assistance from upper extremities and then return to a seated position without upper extremity assist.
Performance Measure- Timed Up and Go Test | 3, 6, 12 and 24 months
  Participants begin in a seated position. They are directed to stand and walk 3 meters to a cone on the floor. They are to round the cone in a continuous motion, walk back to the chair, turn again and be seated. The entire test is performed at a comfortable and safe speed for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Karunakar, MD, Principal Investigator — Wake Forest University Health Sciences; Rachel Seymour, PhD, Study Director — Wake Forest University Health Sciences
Locations (1):
- Atrium Health- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Demetriades D, Karaiskakis M, Toutouzas K, Alo K, Velmahos G, Chan L. Pelvic fractures: epidemiology and predictors of associated abdominal injuries and outcomes. J Am Coll Surg. 2002 Jul;195(1):1-10. doi: 10.1016/s1072-7515(02)01197-3. PMID 12113532
- [Result] Katsoulis E, Giannoudis PV. Impact of timing of pelvic fixation on functional outcome. Injury. 2006 Dec;37(12):1133-42. doi: 10.1016/j.injury.2006.07.017. Epub 2006 Nov 7. PMID 17092504
- [Result] Wong JM, Bucknill A. Fractures of the pelvic ring. Injury. 2017 Apr;48(4):795-802. doi: 10.1016/j.injury.2013.11.021. Epub 2013 Dec 2. PMID 24360668
- [Result] Vallier HA, Cureton BA, Schubeck D. Pelvic ring injury is associated with sexual dysfunction in women. J Orthop Trauma. 2012 May;26(5):308-13. doi: 10.1097/BOT.0b013e31821d700e. PMID 22011632
- [Result] Metze M, Tiemann AH, Josten C. Male sexual dysfunction after pelvic fracture. J Trauma. 2007 Aug;63(2):394-401. doi: 10.1097/01.ta.0000241145.02748.df. PMID 17693842
- [Result] Collinge CA, Archdeacon MT, LeBus G. Saddle-horn injury of the pelvis. The injury, its outcomes, and associated male sexual dysfunction. J Bone Joint Surg Am. 2009 Jul;91(7):1630-6. doi: 10.2106/JBJS.H.00477. PMID 19571085
- [Result] Reilly MC, Zinar DM, Matta JM. Neurologic injuries in pelvic ring fractures. Clin Orthop Relat Res. 1996 Aug;(329):28-36. doi: 10.1097/00003086-199608000-00005. PMID 8769433
- [Result] Suzuki T, Shindo M, Soma K, Minehara H, Nakamura K, Uchino M, Itoman M. Long-term functional outcome after unstable pelvic ring fracture. J Trauma. 2007 Oct;63(4):884-8. doi: 10.1097/01.ta.0000235888.90489.fc. PMID 18090021
- [Result] Tornetta P 3rd, Matta JM. Outcome of operatively treated unstable posterior pelvic ring disruptions. Clin Orthop Relat Res. 1996 Aug;(329):186-93. doi: 10.1097/00003086-199608000-00022. PMID 8769450
- [Result] Pohlemann T, Gansslen A, Schellwald O, Culemann U, Tscherne H. Outcome after pelvic ring injuries. Injury. 1996;27 Suppl 2:B31-8. PMID 8915200
- [Result] Cole JD, Blum DA, Ansel LJ. Outcome after fixation of unstable posterior pelvic ring injuries. Clin Orthop Relat Res. 1996 Aug;(329):160-79. doi: 10.1097/00003086-199608000-00020. PMID 8769448
- [Result] Brenneman FD, Katyal D, Boulanger BR, Tile M, Redelmeier DA. Long-term outcomes in open pelvic fractures. J Trauma. 1997 May;42(5):773-7. doi: 10.1097/00005373-199705000-00003. PMID 9191654
- [Result] Mullis BH, Sagi HC. Minimum 1-year follow-up for patients with vertical shear sacroiliac joint dislocations treated with iliosacral screws: does joint ankylosis or anatomic reduction contribute to functional outcome? J Orthop Trauma. 2008 May-Jun;22(5):293-8. doi: 10.1097/BOT.0b013e31816b6b4e. PMID 18448980
- [Result] Nepola JV, Trenhaile SW, Miranda MA, Butterfield SL, Fredericks DC, Riemer BL. Vertical shear injuries: is there a relationship between residual displacement and functional outcome? J Trauma. 1999 Jun;46(6):1024-9; discussion 1029-30. doi: 10.1097/00005373-199906000-00007. PMID 10372618
- [Result] Dujardin FH, Hossenbaccus M, Duparc F, Biga N, Thomine JM. Long-term functional prognosis of posterior injuries in high-energy pelvic disruption. J Orthop Trauma. 1998 Mar-Apr;12(3):145-50; discussion 150-1. doi: 10.1097/00005131-199803000-00001. PMID 9553853
- [Result] Hoffmann MF, Jones CB, Sietsema DL. Persistent impairment after surgically treated lateral compression pelvic injury. Clin Orthop Relat Res. 2012 Aug;470(8):2161-72. doi: 10.1007/s11999-012-2247-1. PMID 22278851
- [Result] Lefaivre KA, Slobogean G, Starr AJ, Guy P, O'brien PJ, Macadam SA. Methodology and interpretation of radiographic outcomes in surgically treated pelvic fractures: a systematic review. J Orthop Trauma. 2012 Aug;26(8):474-81. doi: 10.1097/BOT.0b013e3182323aa2. PMID 22391403
- [Result] Borg T, Berg P, Fugl-Meyer K, Larsson S. Health-related quality of life and life satisfaction in patients following surgically treated pelvic ring fractures. A prospective observational study with two years follow-up. Injury. 2010 Apr;41(4):400-4. doi: 10.1016/j.injury.2009.11.006. Epub 2009 Dec 14. PMID 20005513
- [Result] Oliver CW, Twaddle B, Agel J, Routt ML Jr. Outcome after pelvic ring fractures: evaluation using the medical outcomes short form SF-36. Injury. 1996 Nov;27(9):635-41. doi: 10.1016/s0020-1383(96)00100-3. PMID 9039360
- [Result] Papakostidis C, Kanakaris NK, Kontakis G, Giannoudis PV. Pelvic ring disruptions: treatment modalities and analysis of outcomes. Int Orthop. 2009 Apr;33(2):329-38. doi: 10.1007/s00264-008-0555-6. Epub 2008 May 7. PMID 18461325
- [Result] Lefaivre KA, Slobogean GP, Valeriote J, O'Brien PJ, Macadam SA. Reporting and interpretation of the functional outcomes after the surgical treatment of disruptions of the pelvic ring: a systematic review. J Bone Joint Surg Br. 2012 Apr;94(4):549-55. doi: 10.1302/0301-620X.94B4.27960. PMID 22434474